CLINICAL TRIAL: NCT00187070
Title: Large Cell Lymphoma, Pilot Study III
Brief Title: Large Cell Lymphoma Pilot Study III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: John T. Sandlund , M.D./Principal Investigator, St.Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCLIII
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Lymphoma, Large Cell; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Non-Hodgkin | interventions — Doxorubicin; Trimethoprim, Sulfamethoxazole Drug Combination; Carboplatin; Ifosfamide; Dexamethasone; Prednisone; Vincristine; Cytarabine; Methotrexate; Etoposide; Cyclophosphamide; Vinblastine; Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Doxorubicin, Cotrimoxazole, Carboplatin, Ifosfamide, Dexamethasone, Prednisone, Vincristine, Cytarabine, Methotrexate, Etoposide, Cyclophosphamide, Vinblastine; Procedure: Stem cell transplant,; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Doxorubicin, Cotrimoxazole, Carboplatin, Ifosfamide, Dexamethasone, Prednisone, Vincristine, Cytarabine, Methotrexate, Etoposide, Cyclophosphamide, Vinblastine — See Detailed Description section for details of treatment interventions.
Procedure: Stem cell transplant, — See Detailed Description section for details of treatment interventions.
Radiation: Radiation Therapy — See Detailed Description section for details of treatment interventions.

SUMMARY:
The main purpose of this study is to find out if it is feasible to deliver a multi-agent chemotherapy regimen which features a shorter, more intensive, immunophenotype-directed approach, and includes an intensification phase with hematopoietic stem cell support for children with large cell lymphoma

DETAILED DESCRIPTION:
Secondary objectives will include documenting the toxicity associated with the treatment regimen, and to estimate the response rates and survival of participants with large cell lymphoma treated on this protocol.

Patients will be treated with induction, consolidation, and maintenance treatment.

Induction

MIED chemotherapy - High dose methotrexate, ifosfamide, etoposide, and dexamethasone for 2 cycles.

High-dose methotrexate 8 gm/m2 on Day 1 with leucovorin rescue Ifosfamide 2 gm/m2/day on days 2-4 (total of 3 days) Etoposide (VP-16) 200 mg/m2/day on Days 2-4 (total of 3 days) Dexamethasone 40 mg/m2/day IV on days 1-4 (given IV or PO daily x 4) Intrathecal MHA, age adjusted dosages.

Consolidation

COPADM chemotherapy for 2 cycles - cyclophosphamide, vincristine, prednisone, adriamycin, high-dose methotrexate

COPAM#1 High dose methotrexate (HD MTX) 5 gm/m2 IV over 4 hours on Day 1 with leucovorin rescue; Doxorubicin 60 mg/m2 IV over 6 hours on Day 2, Vincristine 2.0 mg/m2 (2.0 mg max) Day 1, Cyclophosphamide 500 mg/m2/day (divided every 12 hours) Days 2-4, Prednisone 60 mg/m2 (divided bid) Days 1-5, Intrathecal MHA, age adjusted dosages.

COPADM#2 - like COPADM#1 except: 1. cyclophosphamide dose increased to 1 gm/m2/day divided every 12 hours on Days 2-4, and 2. second dose of vincristine given on Day 6.

DAC chemotherapy x 1 cycle - Dexamethasone, cytarabine, and carboplatin

Carboplatin (AUC of 8) Day 1; Ara-C 2 gm/m2/dose q12 x 2 Day 2 Dexamethasone 40 mg/m2/day Days 1-4; ITMHA dose age adjusted.

Hematopoietic Stem Cell Transplantation - high-dose cyclophosphamide and etoposide

Involved field radiation to the primary tumor will be given over 3-4 weeks. Participants with CNS disease at diagnosis will also receive cranial irradiation.

Maintenance chemotherapy

Vinblastine 6 mg/m2 IV weekly for one year

ELIGIBILITY:
Inclusion Criteria:

* Patient must be previously untreated, except for steroids or emergency radiation therapy.
* Patient must be less than or equal to 18 years of age.
* Patient must have a histologic diagnosis of large cell Non-Hodgkin lymphoma.
* The immunophenotype of tumor cells must be either T-cell or non-B-cell, non-T-cell.

Exclusion Criteria:

* Participants with B-cell immunophenotype NHL.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 1997-12; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
To demonstrate the feasibility of delivery of a multiagent chemotherapy regimen which features a shorter, more direct approach, and includes a phase that incorporates hematopoietic stem cell support for children with large cell lymphoma. | July 2001

CONTACTS AND LOCATIONS:
Overall Officials: John T. Sandlund, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Reaearch Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org